CLINICAL TRIAL: NCT00456495
Title: Effect of Ranibizumab on Malignant Conjunctival Neoplasia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The New York Eye Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Paul T. Finger, MD, Principal Investigator, The New York Eye Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4192s
Record Dates: First submitted 2007-04-03; First posted 2007-04-05 (Estimated); Results first posted 2013-06-06 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-06

CONDITIONS: Conjunctival Neoplasms
MeSH Terms: conditions — Conjunctival Neoplasms | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subconjunctival ranibizumab (Experimental): Patients will receive subconjunctival ranibizumab every 2-4 weeks.
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — Subconjunctival injection of drug every 2 to 4 weeks
  Other Names: Lucentis

SUMMARY:
The purpose of this study is to test the safety and tolerability of subconjunctival injection of ranibizumab in the treatment of malignant conjunctival neoplasia using the incidence and severity of adverse events.

Our secondary objective is to assess the efficacy of ranibizumab treatment on malignant conjunctival neoplasia by evaluating tumor destruction or reduction as documented by slit-lamp photography and ultrasonographic imaging and the regression of blood vessels.

DETAILED DESCRIPTION:
Ranibizumab is a recently approved vascular endothelial growth factor (VEGF) inhibitor shown to be effective in treating exudative macular degeneration. Its analog, Avastin has also been employed to treat macular edema, proliferative diabetic retinopathy and wet age related macular degeneration. Ranibizumab binds to and inhibits vascular endothelial growth factor A (VEGF-A), which has been shown to cause neovascularization and leakage in models of ocular angiogenesis. Binding to VEGF-A prevents ranibizumab's interaction with VEGFR-1 and -2 receptors on the surface of endothelial cells, thereby reducing proliferation, vascular leakage, and angiogenesis.

Given that conjunctival tumors require the formation of new blood vessels to supply the proliferating cells, we propose a study to evaluate the effect of subconjunctival ranibizumab as a primary intervention in patients with conjunctival tumors.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 21 years
* Tumors whose treatment with standard therapy would cause significant visual morbidity
* Diagnosis of biopsy proven malignant conjunctival neoplasia and are
* Recurrent disease
* Multi-focal disease
* Diffuse disease

Exclusion Criteria:

* Extension of tumor into eye or orbit.
* Regional spread or metastatic disease
* Pregnancy (positive pregnancy test) or lactation.
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
* Current infection or inflammation in either eye
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul T. Finger, MD, Principal Investigator — The New York Eye Cancer Center
Locations (1):
- The New York Eye Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Finger PT, Chin KJ. Refractory squamous cell carcinoma of the conjunctiva treated with subconjunctival ranibizumab (Lucentis): a two-year study. Ophthalmic Plast Reconstr Surg. 2012 Mar-Apr;28(2):85-9. doi: 10.1097/IOP.0b013e3182392f29. PMID 22186988

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Five consecutive subjects were enrolled over an 18-month period in a single ophthalmic oncology center.
Pre-assignment Details: There was a single ARM in this study. Subconjunctival 0.5 mg ranibizumab was given as intervention every 2-4 weeks.
Groups:
- Squamous Carcinoma of Conjunctiva: Subconjunctival 0.5 mg ranibizumab
Period: Overall Study
Arm/Group | Squamous Carcinoma of Conjunctiva
Started | 5
Completed | 3
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Squamous Carcinoma of Conjunctiva
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Assessed for Safety and Tolerability
Description: To test the safety and tolerability of subconjunctival injection of ranibizumab in the treatment of malignant conjunctival neoplasia - using comparative slit lamp examination [anterior segment and ocular adnexal examination for adverse events (eg abrasion, melting), visual acuity (number of patients with decrease in visual acuity), and blood pressure at each visit (number of patients with increased blood pressure from baseline), and monthly urinalyis (number of patients with abnormal protein level in urine).
Time Frame: 2 years
Population: Analysis was per protocol. Treatment was delivered every 2-4 weeks with good safety and tolerability
Measure: Number; unit: participants
Groups:
- Open Label Treatment: Patients will receive treatment every 2-4 weeks
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 5
participants | 5

2. Secondary Outcome: Evaluating Tumor Destruction or Reduction
Description: To evaluate the efficacy of treatment using comparative slit lamp examinations (anterior segment and ocular adnexal exam) to evaluate tumor volume, from baseline to month 12, and 24. To report on the number of patients with improvement in tumor volume.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Open Label Treatment: Patients will receive treatment every 2-4 weeks. To evaluate the efficacy of treatment using comparative slit lamp examinations (anterior segment and ocular adnexal exam) to evaluate the number of clock hours of corneal neovascularization, from baseline to month 12, and 24. To report on the number of patients with a decrease in corneal neovascularization.
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 5
Participants | 5

ADVERSE EVENTS:
Time Frame: Monthly over a two year period.
Arm/Group | Squamous Carcinoma of Conjunctiva
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
This was a small case series involving a small number of subjects. Further investigations for dose, drug delivery and case selection are warranted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No